CLINICAL TRIAL: NCT07332559
Title: Effects of Task-oriented Intervention for Pre-handwriting Performance in Preschool Children
Brief Title: Task-Oriented Writing Intervention for Preschoolers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N202312088
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Preschool Child; Handwriting

STUDY DESIGN:
Intervention Model Description: Educational and behavioral intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-Oriented Writing Intervention (Experimental)
  Interventions: Behavioral: Task-Oriented Writing Intervention
- Control group (Active Comparator)
  Interventions: Behavioral: Conventional Fine Motor Training

INTERVENTIONS:
Behavioral: Task-Oriented Writing Intervention — The task-oriented writing intervention consists of structured, goal-directed writing activities designed to support the development of writing performance in preschool children. The intervention focuses on functional writing tasks that are meaningful and relevant to daily learning contexts. Sessions are delivered in a structured educational setting and emphasize active participation and practice.
  Arms: Task-Oriented Writing Intervention
Behavioral: Conventional Fine Motor Training — Participants in the control group receive conventional fine motor training focusing on hand function, coordination, and activities relevant to daily participation, without the task-oriented writing intervention.
  Arms: Control group

SUMMARY:
This study investigates the effectiveness of a task-oriented writing intervention in improving writing performance among preschool children. The intervention is designed to enhance early writing-related abilities through structured, goal-directed writing tasks that reflect functional and meaningful activities.

Eligible preschool children will participate in a series of task-oriented writing sessions delivered in a structured learning environment. Writing performance will be assessed before and after the intervention to examine changes associated with participation in the program.

Findings from this study are expected to provide evidence to support the use of task-oriented writing interventions in early childhood educational and therapeutic settings.

ELIGIBILITY:
Inclusion Criteria: Preschool children diagnosed with sensory integration dysfunction.

Exclusion Criteria:Children who are unable to follow simple instructions required for participation in the intervention.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The Berry-Buktenica Developmental Test of Visual-Motor Integration | Baseline (pre-intervention), immediately post-intervention, and 4 weeks after completion of the intervention
Test of Visual Perceptual Skills-4th Edition | Baseline (pre-intervention), immediately post-intervention, and 4 weeks after completion of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Wan Fang Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No